CLINICAL TRIAL: NCT04064905
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability, and Immunogenicity of Zika Vaccine mRNA-1893 in Healthy Flavivirus Seropositive and Seronegative Adults
Brief Title: Safety, Tolerability, and Immunogenicity of Zika Vaccine mRNA-1893 in Healthy Flavivirus Seropositive and Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1893-P101; BARDA HHS010020160029C (Other Grant/Funding Number: Biomedical Advanced Research & Development Authority (BARDA))
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Zika Virus
Keywords: mRNA-1893; zika vaccine; Moderna
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1893 (Experimental)
  Interventions: Biological: mRNA-1893
- Placebo (Placebo Comparator): 0.9% sodium chloride
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1893 — Zika vaccine
  Arms: mRNA-1893
Other: Placebo — 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
This clinical study will evaluate the safety, tolerability and reactogenicity of mRNA-1893 Zika vaccines in flavivirus seronegative and flavivirus seropositive participants

ELIGIBILITY:
Inclusion Criteria:

* Agrees to comply with the study procedures and provides written informed consent
* 18 to 49 years of age
* In the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., complete diary cards, return for follow-up visits, be available for safety telephone calls).
* Is in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, and physical examination at screening.
* Negative urine pregnancy test at the Screening visit and at the day of each vaccination for females of childbearing potential.
* Male participants must agree to practice adequate contraception from the time of the first vaccination and through 3 months following the last vaccination.
* For flavivirus-seropositive group, has positive flavivirus test results (including dengue, West Nile, and Zika) as determined by enzyme-linked immunosorbent assay (ELISA) or other commercially available serological assay.
* For flavivirus-seronegative group, has negative flavivirus test results (including dengue, West Nile, and Zika) as determined by ELISA or other commercially available serological assay.

Exclusion Criteria:

* Has any acute or chronic, Clinically Significant disease in the opinion of the investigator.
* Has received a vaccine for dengue, Japanese encephalitis, tick-borne encephalitis, West Nile, Yellow Fever, or Zika.
* Has a neurologic disorder
* Has a body mass index that is ≤ 18 or ≥ 35 kg/m2.
* Has elevated liver function tests
* Has clinical laboratory test results (hematology, serum chemistry, or coagulation) with a toxicity score of Grade ≥ 1 at Screening.
* Has a bleeding disorder that would contraindicate IM injections or phlebotomy.
* Reports a diagnosis of congenital or acquired immunodeficiency (including HIV infection), or autoimmune disease.
* Has a history of hypersensitivity or severe reactions to previous vaccinations or any component of the study vaccine.
* Has a history of idiopathic urticaria.
* Reports a previous diagnosis of hematologic malignancy or pre-malignancy or a diagnosis of any other malignancy within the previous 10 years (excluding nonmelanoma skin cancer).
* Has a medical, psychiatric, or occupational condition that, in the opinion of the investigator, might pose an additional risk to the participant due to participation in the study or would interfere with the evaluation of the study vaccines or the interpretation of study results.
* Is acutely ill or febrile on the day of screening (Day 0) or randomization (Day 1).
* Has a history of inflammatory arthritis.
* Has a history of febrile disease with arthritis or arthralgia within 2 weeks of administration of any study vaccine.
* Has received an investigational or nonregistered product (drug or vaccine) within 30 days before the first dose of study vaccine or has plans for administration during the study period.
* Has received or is scheduled to receive an inactivated vaccine within the period from 14 days before, or through 14 days after, administration of any study vaccination.
* Has received or is scheduled to receive a live virus vaccine administered within the period from 28 days before, or through 28 days after, any dose of study vaccine.
* Has received chronic administration (defined as > 14 total days) of immunosuppressants or other immune-modifying drugs within 6 months before the first study vaccine dose.
* Has received immunoglobulins and/or blood products within the 3 months before the first study vaccine dose or has plans for administration during the study period.
* Has a positive test result at the Screening Visit for hepatitis B surface antigen, hepatitis C virus antibody, or HIV type 1 or 2 antibodies.
* Has donated > 450 mL of whole blood or blood products within 30 days of enrollment or plans to do so during the study period.
* Is an immediate family member or household member of study personnel.
* Previously participated in an investigational study involving LNPs.
* Has a positive urine drug screen result at Screening for any of the following nonprescription drugs of abuse: amphetamines, benzodiazepines, cocaine, methadone, opiates, and phencyclidine.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Meridan Clinical Research, Omaha, Nebraska
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
- Ponce School of Medicine - CAIMED Center, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Essink B, Chu L, Seger W, Barranco E, Le Cam N, Bennett H, Faughnan V, Pajon R, Paila YD, Bollman B, Wang S, Dooley J, Kalidindi S, Leav B. The safety and immunogenicity of two Zika virus mRNA vaccine candidates in healthy flavivirus baseline seropositive and seronegative adults: the results of two randomised, placebo-controlled, dose-ranging, phase 1 clinical trials. Lancet Infect Dis. 2023 May;23(5):621-633. doi: 10.1016/S1473-3099(22)00764-2. Epub 2023 Jan 19. PMID 36682364

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to mRNA-1893 by IM injection on Days 1 and 29.
- mRNA-1893 10 mcg: Participants received mRNA-1893 10 mcg by IM injection on Days 1 and 29.
- mRNA-1893 30 mcg: Participants received mRNA-1893 30 mcg by IM injection on Days 1 and 29.
- mRNA-1893 100 mcg: Participants received mRNA-1893 100 mcg by IM injection on Days 1 and 29.
- mRNA-1893 250 mcg: Participants received mRNA-1893 250 mcg by IM injection on Days 1 and 29.
Period: Overall Study
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Started | 24 | 24 | 24 | 24 | 24
Received First Vaccination | 24 | 24 | 24 | 24 | 24
Received Second Vaccination | 24 | 23 | 23 | 24 | 24
Completed | 24 | 21 | 23 | 20 | 22
Not Completed | 0 | 3 | 1 | 4 | 2
Not completed — Lost to Follow-up | 0 | 3 | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all participants who received at least 1 dose of study vaccine (mRNA-1893 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 24 | 24 | 24 | 120
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 11 | 14 | 11 | 70
  Male | 8 | 6 | 13 | 10 | 13 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 8 | 5 | 5 | 29
  Not Hispanic or Latino | 18 | 19 | 16 | 19 | 19 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 2 | 9 | 1 | 12 | 28
  White | 20 | 21 | 14 | 22 | 12 | 89
  Other | 0 | 0 | 1 | 0 | 0 | 1
Flavivirus Serostatus [Count of Participants; unit: Participants]
  Seropositive | 4 | 4 | 4 | 4 | 4 | 20
  Seronegative | 20 | 20 | 20 | 20 | 20 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactogenicity Adverse Reaction (ARs)-First Vaccination
Description: Solicited ARs (local and systemic) were collected in the daily diary. Local ARs included: injection site pain, injection site erythema, and injection site induration/swelling. Systemic ARs included: body temperature (oral), generalized myalgia (muscle ache or pain), generalized arthralgia (joint ache or pain), headache, fatigue/malaise (unusual tiredness), nausea/vomiting, chills, and rash. Data for this outcome measure is reported up to 7 days after the first study vaccination only. A summary of all serious adverse events (SAEs) and all nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: Up to Day 7 after first vaccination (up to 8 days)
Population: The First Vaccination Solicited Safety Set consisted of all participants in the Safety Set who had received the first study vaccination and had contributed any solicited AR data (local or systemic reactogenicity events) from the time of first study vaccination through the following 7 days. Here, number analyzed signifies those participants who were evaluable at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 24 | 24 | 23 | 24 | 24
Participants
  Local ARs- Erythema (Redness): number analyzed (Participants) | 22 | 24 | 21 | 24 | 22
  Local ARs- Erythema (Redness) | 0 | 0 | 0 | 1 | 2
  Local ARs- Pain: number analyzed (Participants) | 23 | 24 | 23 | 24 | 24
  Local ARs- Pain | 1 | 12 | 12 | 17 | 14
  Local ARs- Swelling (Hardness): number analyzed (Participants) | 22 | 24 | 21 | 24 | 22
  Local ARs- Swelling (Hardness) | 0 | 0 | 0 | 0 | 1
  Systemic ARs- Arthralgia: number analyzed (Participants) | 22 | 24 | 23 | 24 | 24
  Systemic ARs- Arthralgia | 1 | 2 | 2 | 0 | 1
  Systemic ARs- Chills: number analyzed (Participants) | 22 | 24 | 23 | 24 | 24
  Systemic ARs- Chills | 0 | 1 | 0 | 0 | 2
  Systemic ARs- Fatigue: number analyzed (Participants) | 22 | 24 | 23 | 24 | 24
  Systemic ARs- Fatigue | 3 | 8 | 5 | 3 | 4
  Systemic ARs- Fever | 0 | 1 | 0 | 1 | 0
  Systemic ARs- Headache: number analyzed (Participants) | 22 | 24 | 23 | 24 | 24
  Systemic ARs- Headache | 4 | 7 | 5 | 3 | 3
  Systemic ARs- Myalgia: number analyzed (Participants) | 22 | 24 | 23 | 24 | 24
  Systemic ARs- Myalgia | 2 | 5 | 3 | 1 | 6
  Systemic ARs- Nausea: number analyzed (Participants) | 22 | 24 | 23 | 24 | 24
  Systemic ARs- Nausea | 0 | 4 | 3 | 3 | 0
  Systemic ARs- Rash | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactogenicity Adverse Reaction (ARs)-Second Vaccination
Description: Solicited ARs (local and systemic) were collected in the daily diary. Local ARs included: injection site pain, injection site erythema, and injection site induration/swelling. Systemic ARs included: body temperature (oral), generalized myalgia (muscle ache or pain), generalized arthralgia (joint ache or pain), headache, fatigue/malaise (unusual tiredness), nausea/vomiting, chills, and rash. Data for this outcome measure is reported up to 7 days after the second study vaccination only. A summary of all serious adverse events (SAEs) and all nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: Up to Day 7 after second vaccination (Day 29 to Day 36)
Population: The Second Vaccination Solicited Safety Set consisted of all participants in the Safety Set who had received the second study vaccination and had contributed any solicited AR data (local or systemic reactogenicity events) from the time of first study vaccination through the following 7 days. Here, number analyzed signifies those participants who were evaluable at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 23 | 23 | 22 | 24 | 23
Participants
  Local ARs- Erythema (Redness): number analyzed (Participants) | 22 | 23 | 20 | 24 | 23
  Local ARs- Erythema (Redness) | 0 | 0 | 1 | 2 | 2
  Local ARs- Pain: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Local ARs- Pain | 2 | 8 | 11 | 15 | 14
  Local ARs- Swelling (Hardness): number analyzed (Participants) | 22 | 23 | 20 | 24 | 23
  Local ARs- Swelling (Hardness) | 0 | 0 | 2 | 1 | 3
  Systemic ARs- Arthralgia: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Arthralgia | 2 | 4 | 4 | 9 | 7
  Systemic ARs- Chills: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Chills | 3 | 1 | 5 | 11 | 14
  Systemic ARs- Fatigue: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Fatigue | 3 | 6 | 10 | 10 | 13
  Systemic ARs- Fever | 1 | 1 | 3 | 7 | 11
  Systemic ARs- Headache: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Headache | 4 | 5 | 8 | 9 | 13
  Systemic ARs- Myalgia: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Myalgia | 1 | 7 | 4 | 10 | 15
  Systemic ARs- Nausea: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Nausea | 2 | 2 | 1 | 4 | 5
  Systemic ARs- Rash: number analyzed (Participants) | 22 | 23 | 22 | 24 | 23
  Systemic ARs- Rash | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A treatment-emergent adverse event (TEAE) was as any AE not present before exposure to vaccine or any AE already present that worsened in intensity or frequency after exposure. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to Day 392 (all AEs considered an SAE were collected till end of study [Day 392]; the Other AEs [non-SAE] were collected up to Day 57)
Population: The Safety Set consisted of all participants who received at least 1 dose of study vaccine (mRNA-1893 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Participants | 14 | 12 | 13 | 15 | 10

4. Primary Outcome: Number of Participants With Adverse Event of Special Interest (AESI) and Serious Adverse Events (SAEs)
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions was a congenital anomaly/birth defect, or was an important medical event. AESIs included potentially immune-mediated medical conditions (autoimmune or autoinflammatory diseases) that may have the theoretical potential for association with novel vaccines. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Day 1 to the end of study visit (up to Day 392)
Population: The Safety Set consisted of all participants who received at least 1 dose of study vaccine (mRNA-1893 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Participants
  SAEs | 3 | 0 | 0 | 0 | 1
  AESI | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Geometric Mean Titer (GMT) of Neutralizing Antibody (nAb) Against Zika Virus as Measured by Plaque Reduction Neutralization Test (PRNT50)
Description: GMT 95% CI is calculated based on the t-distribution of the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Day 1, 29, 57, Month 7 and 13
Population: Per-Protocol Set consisted of all participants who did not had a major protocol deviation, received vaccine within the acceptable vaccination window and received full dose of assigned vaccine, had immunogenicity samples taken within acceptable visit windows, had a pre-vaccination and the corresponding 1 post-vaccination serum sample available for testing. Here, number analyzed signifies those participants were evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 24 | 24 | 23 | 24 | 24
Titer
  Day 1 | 9.1 [7.0 to 11.8] | 10.1 [7.2 to 14.1] | 8.9 [7.1 to 11.3] | 9.1 [7.0 to 11.9] | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated.
  Day 29 | 9.1 [6.9 to 12.0] | 13.6 [7.8 to 23.8] | 19.8 [11.5 to 33.8] | 54.6 [29.4 to 101.3] | 29.2 [17.2 to 49.3]
  Day 57: number analyzed (Participants) | 23 | 22 | 22 | 24 | 23
  Day 57 | 9.3 [6.8 to 12.5] | 200.5 [121.1 to 331.9] | 267.2 [161.6 to 441.8] | 393.0 [273.1 to 565.7] | 230.0 [148.9 to 355.3]
  Month 7: number analyzed (Participants) | 24 | 21 | 22 | 21 | 23
  Month 7 | 8.9 [7.1 to 11.1] | 42.7 [23.0 to 79.3] | 68.0 [39.7 to 116.3] | 174.8 [114.6 to 266.7] | 116.7 [75.4 to 180.6]
  Month 13: number analyzed (Participants) | 24 | 20 | 21 | 17 | 21
  Month 13 | 9.0 [7.1 to 11.4] | 41.0 [21.7 to 77.4] | 47.8 [23.9 to 95.6] | 100.8 [56.3 to 180.4] | 100.2 [64.5 to 155.7]

6. Secondary Outcome: Geometric Mean Titer of Neutralizing Antibody in Initially Seronegative Participants Against Zika Virus as Measured by Plaque Reduction Neutralization Test (PRNT50)
Description: as for outcome 5
Time Frame: Day 1, 29, 57, Month 7 and 13
Population: Per-Protocol Set: All participants who did not had a major protocol deviation, received vaccine within acceptable vaccination window and received full dose of assigned vaccine, had immunogenicity samples taken within acceptable visit windows, had a pre-vaccination and the corresponding 1 post-vaccination serum sample available for testing. Number of participants analyzed signifies who were evaluable for this endpoint and number analyzed signifies who were evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20
Titer
  Day 1 | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated.
  Day 29 | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 8.5 [7.5 to 9.5] | 14.4 [9.9 to 21.0] | 45.9 [23.4 to 89.9] | 27.6 [15.5 to 49.2]
  Day 57: number analyzed (Participants) | 19 | 18 | 18 | 20 | 19
  Day 57 | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 195.6 [108.4 to 352.8] | 303.4 [195.5 to 470.9] | 454.2 [333.0 to 619.6] | 273.6 [195.3 to 383.2]
  Month 7: number analyzed (Participants) | 20 | 17 | 18 | 17 | 19
  Month 7 | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 38.2 [20.0 to 73.0] | 66.7 [38.5 to 115.4] | 170.1 [112.1 to 258.0] | 137.7 [94.6 to 200.5]
  Month 13: number analyzed (Participants) | 20 | 16 | 17 | 14 | 17
  Month 13 | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated. | 35.0 [18.4 to 66.5] | 48.3 [23.0 to 101.7] | 112.3 [63.6 to 198.4] | 113.2 [77.7 to 164.9]

7. Secondary Outcome: Geometric Mean Titer of Neutralizing Antibody in Initially Seropositive Participants Against Zika Virus as Measured by Plaque Reduction Neutralization Test (PRNT50)
Description: as for outcome 5
Time Frame: Day 1, 29, 57, Month 7 and 13
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Titer
  Day 1 | 17.0 [1.5 to 188.2] | 32.2 [2.5 to 417.7] | 15.2 [2.0 to 115.7] | 17.4 [1.5 to 203.9] | 8.0 [NA to NA] — All values were equal to 8.0, therefore CI (upper and lower limit) could not be calculated.
  Day 29 | 17.8 [1.4 to 226.8] | 147.9 [6.2 to 3507.8] | 88.1 [3.6 to 2166.7] | 130.6 [13.0 to 1306.4] | 38.2 [3.7 to 398.6]
  Day 57 | 18.6 [1.3 to 270.5] | 224.1 [43.5 to 1153.5] | 150.9 [6.2 to 3699.1] | 190.5 [19.2 to 1887.2] | 100.9 [5.4 to 1886.3]
  Month 7 | 15.2 [2.0 to 116.9] | 68.8 [3.6 to 1231.4] | 74.2 [4.0 to 1362.9] | 196.3 [18.3 to 2102.4] | 53.2 [3.7 to 774.9]
  Month 13: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4
  Month 13 | 15.9 [1.8 to 142.9] | 77.6 [3.6 to 1670.2] | 45.6 [1.7 to 1237.6] | 60.9 [0.6 to 6248.0] | 59.6 [3.9 to 922.0]

8. Secondary Outcome: Percentage of Participants Who Seroconverted From Day 1 (Baseline) to Day 29, From Day 1 to Day 57, From Day 1 to Month 7, and From Day 1 to Month 13
Description: Seroconversion is defined as a change of PRNT from below the lower limit of quantification (LLOQ) to a PRNT equal to or above LLOQ for the assay, or a multiplication by at least 4 in participants with pre-existing PRNT titers.
Time Frame: Day 1 (baseline) to Day 29, from Day 1 to Day 57, from Day 1 to Month 7, and from Day 1 to Month 13.
Population: Per-Protocol Set consisted of all participants who did not had a major protocol deviation, received vaccine within the acceptable vaccination window and received full dose of assigned vaccine, had immunogenicity samples taken within acceptable visit windows, had a pre-vaccination and the corresponding 1 post-vaccination serum sample available for testing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 24 | 24 | 23 | 24 | 24
percentage of participants
  Day 1 (baseline) to Day 29 | 0 | 12.5 | 47.8 | 75.0 | 66.7
  Day 1 to Day 57 | 0 | 90.9 | 95.5 | 100.0 | 95.7
  Day 1 to Month 7 | 0 | 66.7 | 81.8 | 100.0 | 95.7
  Day 1 to Month 13 | 0 | 60.0 | 61.9 | 94.1 | 95.2

9. Secondary Outcome: Number of Initially Seronegative Participants With a Seroresponse as Measured by Plaque Reduction Neutralization Test
Description: Seroconversion is defined as a change of PRNT from below the LLOQ to a PRNT equal to or above LLOQ for the assay, or a multiplication by at least 4 in participants with pre-existing PRNT titers.
Time Frame: Day 29, Day 57, Month 7, and Month 13
Population: Per-Protocol Set: All participants who did not had a major protocol deviation, received vaccine within the acceptable vaccination window and received full dose of assigned vaccine, had immunogenicity samples taken within acceptable visit windows, had a pre-vaccination and the corresponding 1 post-vaccination serum sample available for testing. Number of participants analyzed signifies who were evaluable for this endpoint and number analyzed signifies who were evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20
Participants
  Day 29 | 0 | 1 | 8 | 14 | 13
  Day 57 | 0 | 17 | 18 | 20 | 19
  Month 7 | 0 | 12 | 15 | 17 | 19
  Month 13 | 0 | 10 | 11 | 14 | 17

10. Secondary Outcome: Number of Initially Seropositive Participants With a 2-fold or 4-fold Increase in Neutralizing Antibody Titers as Compared With Baseline as Measured by Plaque Reduction Neutralization Test
Description: Seroconversion is defined as a change of Plaque Reduction Neutralization Test from below the lower limit of quantification (LLOQ) to a PRNT equal to or above LLOQ for the assay, or a multiplication by at least 4 in participants with pre-existing PRNT titers.
Time Frame: Day 29, Day 57, Month 7, and Month 13
Population: Per-Protocol Set consisted of all participants who did not had a major protocol deviation, received vaccine within the acceptable vaccination window and received full dose of assigned vaccine, had immunogenicity samples taken within acceptable visit windows, had a pre-vaccination and the corresponding 1 post-vaccination serum sample available for testing. Here, Number of participants analyzed signifies those participants who were evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants
  Day 29: >= 2-fold increase | 0 | 3 | 3 | 3 | 2
  Day 29: >= 4-fold increase | 0 | 2 | 2 | 3 | 2
  Day 57: >= 2-fold increase | 0 | 4 | 3 | 3 | 3
  Day 57: >= 4-fold increase | 0 | 3 | 3 | 3 | 3
  Month 7: >= 2-fold increase | 0 | 2 | 3 | 3 | 2
  Month 7: >= 4-fold increase | 0 | 1 | 2 | 3 | 2
  Month 13: >= 2-fold increase | 0 | 2 | 2 | 2 | 2
  Month 13: >= 4-fold increase | 0 | 1 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Day 1 to the end of study visit (up to Day 392)
Description: The Safety Set consisted of all participants who received at least 1 dose of study vaccine (mRNA-1893 or placebo). Adverse Events reported in the Adverse Events section below include unsolicited AEs and solicited ARs. All AEs considered as an SAE were collected till end of study (Day 392). The Other AEs (non-SAE) were collected up to Day 57.
Arm/Group | Placebo | mRNA-1893 10 mcg | mRNA-1893 30 mcg | mRNA-1893 100 mcg | mRNA-1893 250 mcg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24 | 0/24 | 0/24 | 0/24 | 1/24
Other Adverse Events (participants affected / at risk) | 17/24 | 21/24 | 21/24 | 22/24 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | mRNA-1893 10 mcg (N=24) | mRNA-1893 30 mcg (N=24) | mRNA-1893 100 mcg (N=24) | mRNA-1893 250 mcg (N=24)
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | mRNA-1893 10 mcg (N=24) | mRNA-1893 30 mcg (N=24) | mRNA-1893 100 mcg (N=24) | mRNA-1893 250 mcg (N=24)
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mycoplasma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otosalpingitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nipple infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 8 | 12 | 12 | 11 | 13
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 3 | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 12 | 7 | 11 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 5 | 9 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 3 | 14 | 16 | 20 | 17
Fatigue (General disorders) | 5 | 9 | 11 | 11 | 14
Chills (General disorders) | 3 | 2 | 6 | 11 | 14
Pyrexia (General disorders) | 1 | 2 | 4 | 8 | 11
Injection site erythema (General disorders) | 0 | 0 | 1 | 3 | 3
Injection site swelling (General disorders) | 0 | 0 | 2 | 2 | 3
Infusion site rash (General disorders) | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 2 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT04064905/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT04064905/SAP_001.pdf
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04064905/ICF_002.pdf